CLINICAL TRIAL: NCT03657732
Title: A Multi-center Longitudinal Cohort Study of Familial Alzheimer's Disease in China
Brief Title: The Chinese Familial Alzheimer's Network
Acronym: CFAN
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Chao Yang Hospital (Other); Fu Xing Hospital, Capital Medical University (Other); Peking Union Medical College Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Chinese PLA General Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Geriatric Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Fujian Medical University Union Hospital (Other); Guangzhou Psychiatric Hospital (Other Government); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Handan Central Hospital (Other); Hebei General Hospital (Other); First Hospital of Shijiazhuang City (Other); Tangshan Worker's Hospital (Other); Henan Provincial People's Hospital (Other); Kaifeng Central Hospital (Other); People's Hospital of Zhengzhou University (Other); First Affiliated Hospital of Harbin Medical University (Other); Tongji Hospital (Other); People's Hospital Affiliated Hubei Medical University (Unknown); Zhongnan Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Xiangya Hospital of Central South University (Other); The First Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other); Subei People's Hospital of Jiangsu (Unknown); Nantong University Affiliated Hospital (Unknown); Mineral General Hospital, Xuzhou (Unknown); Jiangxi Provincial People's Hopital (Other); Anshan Central Hospital (Other); Affiliated Zhongshan Hospital of Dalian University (Other); First Hospital of China Medical University (Other); Baotou Central Hospital (Other); General Hospital of Ningxia Medical University (Other); The People's Hospital of Ningxia (Other); The Affiliated Hospital of Qingdao University (Other); The 960th Hospital of PLA (Unknown); Qilu Hospital of Shandong University (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Shandong Provincial Hospital (Other Government); Qingdao Municipal Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Tang-Du Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Ruijin Hospital (Other); RenJi Hospital (Other); Shanghai Changzheng Hospital (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Tianjin Huanhu Hospital (Other); Tianjin Medical University General Hospital (Other); Traditional Chinese Medicine Hospital of Xinjiang Autonomous Region (Unknown); Ningbo Medical Center Lihuili Hospital (Other Government); First Affiliated Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Zhejiang University (Other); Shao Yifu Hospital of Zhejiang Medical University (Unknown); Zhejiang Provincial People's Hospital (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); People's Hospital of Chongqing (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other); Zigong No.1 Peoples Hospital (Other)
Responsible Party: Principal Investigator, Jianping Jia, Chief Director, Capital Medical University
Other Study IDs: SYXWJ002
Record Dates: First submitted 2018-08-21; First posted 2018-09-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease; Familial Alzheimer Disease (FAD)
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Blood, cerebral spinal fluid, saliva, and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Familial Alzheimer's disease group: Familial Alzheimer's disease with the known mutation presenilin1 (PSEN1), presenilin2 (PSEN2) and amyloid precursor protein (APP) including mutation carriers and noncarriers, presymptomatic and symptomatic.
- Normal control group: Normal cognitive control people

SUMMARY:
This research will establish and continuously improve the FAD research network in conjunction with multi-center institutions nationwide. By collecting information on the family's demography, genetics, neuropsychology, neuroimaging, biomarkers and other information, we can understand the current FAD population in China, clarify the genetic characteristics, pathogenesis, disease characteristics and diagnosis and treatment status of AD in China; which will lay the foundation for ameliorating clinical diagnosis and treatment, establishing a Chinese FAD clinical database and an international cooperative research platform.

1. To set up a multi-center, nationwide FAD research network and database platform in China
2. To clarify the epidemiological characteristics of FAD in China.
3. To clarify the genetic characteristics of FAD in China.
4. To clarify the clinical characteristics and disease development laws of FAD.
5. To discover and verify the early diagnosis biomarkers of AD.
6. To establish a genetic counseling model.

DETAILED DESCRIPTION:
1. The network and database include ADAD cohort of the known mutations of PSEN1, PSEN2 and APP (mutation carriers and noncarriers; pre-symptomatic and symptomatic) and unknown mutations cohort.
2. Conduct a comprehensive FAD epidemiological survey in China to clarify the impact of different nationalities, regions, gender, age, living environment (rural/urban), education level, etc. on the occurrence and development of the disease.
3. This project is to discover new FAD mutation sites，pathogenic genes, to protective genes, to explore the pathogenic and protective mechanism, to analyze the disease development laws of families with different sizes of FAD in China, and to clarify the frequency distribution of mutant genes in the Chinese FAD population.
4. The project will collect and regularly follow-up the samples (blood, urine and saliva etc.) and data (neuropsychology, imaging etc.) in the cohort. Emphasis is placed on the occurrence and development of asymptomatic mutant gene carriers from asymptomatic to symptomatic periods.
5. In the FAD family cohort, we will screen high-sensitivity and high-specificity body fluid markers suitable for Chinese people, verify in the SAD cohort, and establish a prediction model of body fluid markers for AD occurrence and disease progression; use structural MRI, dual tracer 18F-FDG PET and 11C-PIB PET multimodal imaging technology, dynamically monitor the dynamic evolution of imaging biomarkers such as brain structure, glucose metabolism and Aβ deposition at various stages of AD progression.
6. We will combine with the genetic characteristics of Chinese FAD to analyze the impact of lifestyle, physical exercise, nootropic drugs, cognitive training, etc. on the disease progression of FAD patients or asymptomatic mutant gene carriers, to establish a genetic counseling model.

ELIGIBILITY:
Familial Alzheimer's disease group

Inclusion criteria:

1. Written informed consent obtained from the participant or a legal guardian prior to any study-related procedures;
2. At least two first-degree relatives in a family have AD (clinically or by testing)，and at least 3 out of 2 generations are patients;
3. At least one family member with normal cognitive function (the age should be greater than the average age of onset of the family);
4. Pedigrees carrying FAD pathogenic genes (APP/PSEN1/PSEN2);
5. People in this family >18 years old can be recruited;
6. Participant is cognitively normal or demented but not reaching bedridden level;
7. Participants are able to provide two reliable informants who can provide clinical information;
8. Dementia is diagnosed according to the criteria described by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-R );
9. The diagnosis of AD is made using the National Institute of Neurologic and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA ) or National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria ;
10. The diagnosis of MCI is made according to Petersen criteria and the classiﬁcation is according to the method of Lopez et al.

Exclusion criteria:

1. Dementia caused by other factors such as depression, other psychiatric illnesses, thyroid dysfunction, encephalitis, multiple sclerosis, brain trauma, brain tumor, syphilis, acquired immunodeficiency syndrome (AIDS), Creutzfeldt-Jakob disease and other types of dementias such as vascular dementia (VaD), frontotemporal dementia (FTD), dementia with Lewy bodies (DLB), and Parkinson's dementia (PDD)；
2. MRI and laboratory tests do not support or rule out a diagnosis of AD；
3. Severe circulatory, respiratory, urinary, digestive, hematopoietic diseases (such as unstable angina, uncontrollable asthma, active gastric bleeding) and cancer；
4. Participant has severe psychiatric illness or severe dementia that would interfere in completing initial and follow-up clinical assessments；
5. Participant has a history of alcoholism or drug abuse；
6. Pregnant or lactating women；
7. No reliable informant；
8. Lumbar puncture exclusion criteria：coagulation disorders or platelet counts < 100,000 cells/μL, lumbar surgery within the last 6 months prior to lumbar puncture that interferes with anatomy of the inter-vertebral spaces, History of chronic or repeated CSF leakage following previous LP(s);
9. MRI Exclusion Criteria: electronic and magnetic metal implants such as pacemakers, artificial heart valve, metal prosthesis, metal joint, etc.; metallic foreign body in the eye; aneurysm clips in the brain.

Normal control group

Inclusion criteria:

1. Aged 18 (inclusive) or above;
2. Normal MMSE and MoCA evaluations. MMSE>19 points for illiteracy, >24 points for those educated less than 7 years, >27 points for those educated equal to or more than 7 years. MoCA>13 points for illiteracy, >19 points for those educated less than 7 years, >24 points for those educated equal to or more than 7 years.

Exclusion criteria:

1. Subjects with abnormal MMSE or MoCA scores;
2. Subjects with a history of cerebral infarction, traumatic brain injury or related manifestations in MRI;
3. Other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.);
4. Other systemic diseases that can cause cognitive impairment (such as liver, renal and thyroid insufficiency, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.);
5. Mental and neurodevelopmental retardation;
6. Suffering from a disease that cannot be combined with a cognitive examination;
7. Contraindications to MRI;
8. Refuse to draw blood;
9. Refuse to sign the informed consent at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with family histroy of Alzheimer's disease, characterised with at least two first-degree relatives.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2005-01-10 (Actual); Primary Completion 2038-01-01 (Estimated); Study Completion 2038-01-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of gene mutations in familial Alzheimer's disease in China. | An Average of 1 year
  Gene analysis of known mutations (PSEN1, PSEN2 and APP), apolipoprotein E (APOE) genotype and unknown mutations in familial Alzheimer's disease patients.
The development patterns of genetic, biofluid, imaging, and neuropsychological markers of FAD. | An Average of 3 to 10 years
  The development patterns of genetic, biofluid, imaging, and neuropsychological markers of FAD. The dynamic changes of biochemical, pathological, structural and functional markers with disease progression.

SECONDARY OUTCOMES:
Changes of neuropsychological function in pedigree members at different stage of cognitive impairment in familial Alzheimer's disease in China. | An Average of 1 year
  Changes of neuropsychological function measured by neuropsychological assessment battery.
Changes of brain structure in pedigree members at different stage of cognitive impairment in familial Alzheimer's disease in China. | An Average of 1 year
  Changes of structure of the whole brain, hippocampus other brain structures measured by MRI.
Changes of brain glucose metabolism in pedigree members at different stage of cognitive impairment in familial Alzheimer's disease in China. | An Average of 1 year
  Changes of glucose metabolism of the whole brain, hippocampus and other brain structures as measured by 18F-fluorodeoxyglucose (FDG)-positron emission tomography (PET).
Changes of brain amyloid deposition in pedigree members at different stage of cognitive impairment in familial Alzheimer's disease in China. | An Average of 1 year
  Changes of amyloid deposition of the whole brain, hippocampus and other brain structures as measured by amyloid PET.
Changes of brain tau deposition in pedigree members at different stage of cognitive impairment in familial Alzheimer's disease in China. | An Average of 1 year
  Changes of tau deposition of the whole brain, hippocampus and other brain structures as measured by tau PET.
Changes of humoral biomarkers in pedigree members at different stage of cognitive impairment in familial Alzheimer's disease in China. | Each biomarker with time frame of average 1 year
  Humoral biomarkers are included Aβ42, Aβ40, phosphated tau and total tau in plasma, cerebrospinal fluid, saliva, and urine.
The effective non-pharmacologic treatment(NPT) intervention | An Average of 1 year
  The effective non-pharmacologic treatment(NPT) intervention- including lifestyle(diet and sleep habits, smoking, drinking and social networking), health products, exercise habits, cognitive training, risk factor control- on APOE ε4 carriers, MCI and dementia patients using questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Jia, Doctor, Study Chair — Xuanwu Hospital of Capital Medical University
Locations (65):
- China (65):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Geriatric Hospital, Changping, Beijing Municipality
  - Beijing Chao Yang Hospital, Chaoyang, Beijing Municipality
  - China-Japan Friendship Hospital, Chaoyang, Beijing Municipality
  - Dongfang Hospital Affiliated to Beijing University of Chinese Medicine, Fengtai, Beijing Municipality
  - Chinese PLA General Hospital, Haidian, Beijing Municipality
  - Fu Xing Hospital, Capital Medical University, Haidian, Beijing Municipality
  - Peking University Third Hospital, Haidian, Beijing Municipality
  - Peking Union Medical College Hospital, Xicheng, Beijing Municipality
  - Peking University First Hospital, Xicheng, Beijing Municipality
  - Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Yuzhong, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Yuzhong, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fujian, Guangdong
  - Guangzhou Psychiatric Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Zhongshan, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital Of Guizhou Medical University, Guiyang, Guizhou
  - Handan Central Hospital, Handan, Hebei
  - First Hospital of Shijiazhuang City, Shijiazhuang, Hebei
  - Tangshan Worker's Hospital, Tangshan, Hebei
  - Hebei General Hospital, Zhijiazhuang, Hebei
  - First Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - People's Hospital Affiliated Hubei Medical University, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Wuhan, Hunan
  - Wuhan University Zhongnan Hospital, Wuhan, Hunan
  - Xiangya Hospital of Central South University, Wuhan, Hunan
  - Nantong University Affiliated Hospital, Nantong, Jiangsu
  - Subei People's Hospital of Jiangsu, Subei, Jiangsu
  - Mineral General Hospital, Xuzhou, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - China-Japan friendship Hospital of Jilin university, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Changda Hospital, Anshan, Anshan, Liaoning
  - Affiliated Zhongshan hospital of Dalian university, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - First Hospital of China Medical University, Shenyang, Liaoning
  - Baotou Central Hospital, Baotou, Nei Monggol
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The People's Hospital of Ningxia, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jining, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao, Shandong
  - QingDao Municipal Hospital, Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The 88th Hospital of PLA, Tai’an, Shandong
  - Shanghai Changzheng Hospital, Huangpu, Shanghai Municipality
  - Ruijin Hospital, Luwan, Shanghai Municipality
  - RenJi Hospital, Putong, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - First Affiliated Hospital Xi'an Jiaotong University, Xi’an, Shanxi
  - Tang-Du Hospital, Xi’an, Shanxi
  - Afﬁliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Zigong First People's Hospital, Zigong, Sichuan
  - Tianjin Huanhu Hospital, Xianshuigu, Tianjin Municipality
  - Tianjin Medical University General Hospital, Xiaobailou, Tianjin Municipality
  - Traditional Chinese Medicine Hospital of Xinjiang Autonomous Region, Ürümqi, Xinjiang
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Shao Yifu Hospital of Zhejiang Medical University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo City Medical Treatment Center Lihuili Hospital, Ningbo, Zhejiang
  - First Affiliated Hospital of Wenzhou Medical Univeristy, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yang H, Hou T, Wang W, Luo Y, Yan F, Jia J. The Effect of Chronic Cerebral Hypoperfusion on Amyloid-beta Metabolism in a Transgenic Mouse Model of Alzheimer's Disease (PS1V97L). J Alzheimers Dis. 2018;62(4):1609-1621. doi: 10.3233/JAD-171094. PMID 29614686
- [Result] Hou TT, Yang HY, Wang W, Wu QQ, Tian YR, Jia JP. Sulforaphane Inhibits the Generation of Amyloid-beta Oligomer and Promotes Spatial Learning and Memory in Alzheimer's Disease (PS1V97L) Transgenic Mice. J Alzheimers Dis. 2018;62(4):1803-1813. doi: 10.3233/JAD-171110. PMID 29614663
- [Result] Wang Q, Jia J, Qin W, Wu L, Li D, Wang Q, Li H. A Novel AbetaPP M722K Mutation Affects Amyloid-beta Secretion and Tau Phosphorylation and May Cause Early-Onset Familial Alzheimer's Disease in Chinese Individuals. J Alzheimers Dis. 2015;47(1):157-65. doi: 10.3233/JAD-143231. PMID 26402764
- [Result] Jia J, Zuo X, Jia XF, Chu C, Wu L, Zhou A, Wei C, Tang Y, Li D, Qin W, Song H, Ma Q, Li J, Sun Y, Min B, Xue S, Xu E, Yuan Q, Wang M, Huang X, Fan C, Liu J, Ren Y, Jia Q, Wang Q, Jiao L, Xing Y, Wu X; China Cognition and Aging Study (China COAST) Group. Diagnosis and treatment of dementia in neurology outpatient departments of general hospitals in China. Alzheimers Dement. 2016 Apr;12(4):446-53. doi: 10.1016/j.jalz.2015.06.1892. Epub 2015 Aug 7. PMID 26256457
- [Result] Wang W, Lu L, Wu QQ, Jia JP. Brain Amyloid-beta Plays an Initiating Role in the Pathophysiological Process of the PS1V97L-Tg Mouse Model of Alzheimer's Disease. J Alzheimers Dis. 2016 Apr 12;52(3):1089-99. doi: 10.3233/JAD-160004. PMID 27079718
- [Result] Dong J, Qin W, Wei C, Tang Y, Wang Q, Jia J. A Novel PSEN1 K311R Mutation Discovered in Chinese Families with Late-Onset Alzheimer's Disease Affects Amyloid-beta Production and Tau Phosphorylation. J Alzheimers Dis. 2017;57(2):613-623. doi: 10.3233/JAD-161188. PMID 28269784
- [Result] Zhang G, Xie Y, Wang W, Feng X, Jia J. Clinical characterization of an APP mutation (V717I) in five Han Chinese families with early-onset Alzheimer's disease. J Neurol Sci. 2017 Jan 15;372:379-386. doi: 10.1016/j.jns.2016.10.039. Epub 2016 Oct 28. PMID 27838006
- [Result] Wang Y, Cheng Z, Qin W, Jia J. Val97Leu mutant presenilin-1 induces tau hyperphosphorylation and spatial memory deficit in mice and the underlying mechanisms. J Neurochem. 2012 Apr;121(1):135-45. doi: 10.1111/j.1471-4159.2011.07489.x. Epub 2012 Feb 10. PMID 21929538
- [Result] Qin W, Jia J. Down-regulation of insulin-degrading enzyme by presenilin 1 V97L mutant potentially underlies increased levels of amyloid beta 42. Eur J Neurosci. 2008 May;27(9):2425-32. doi: 10.1111/j.1460-9568.2008.06207.x. PMID 18445230
- [Result] Fang B, Jia L, Jia J. Chinese Presenilin-1 V97L mutation enhanced Abeta42 levels in SH-SY5Y neuroblastoma cells. Neurosci Lett. 2006 Oct 2;406(1-2):33-7. doi: 10.1016/j.neulet.2006.06.072. Epub 2006 Aug 17. PMID 16916581
- [Result] Jia J, Xu E, Shao Y, Jia J, Sun Y, Li D. One novel presenilin-1 gene mutation in a Chinese pedigree of familial Alzheimer's disease. J Alzheimers Dis. 2005 Apr;7(2):119-24; discussion 173-80. doi: 10.3233/jad-2005-7204. PMID 15851849
- [Result] Jia L, Xu H, Chen S, Wang X, Yang J, Gong M, Wei C, Tang Y, Qu Q, Chu L, Shen L, Zhou C, Wang Q, Zhao T, Zhou A, Li Y, Li F, Li Y, Jin H, Qin Q, Jiao H, Li Y, Zhang H, Lyu D, Shi Y, Song Y, Jia J. The APOE epsilon4 exerts differential effects on familial and other subtypes of Alzheimer's disease. Alzheimers Dement. 2020 Dec;16(12):1613-1623. doi: 10.1002/alz.12153. Epub 2020 Sep 3. PMID 32881347
- [Result] Quan M, Zhao T, Tang Y, Luo P, Wang W, Qin Q, Li T, Wang Q, Fang J, Jia J. Effects of gene mutation and disease progression on representative neural circuits in familial Alzheimer's disease. Alzheimers Res Ther. 2020 Jan 14;12(1):14. doi: 10.1186/s13195-019-0572-2. PMID 31937364
- [Result] Jia L, Fu Y, Shen L, Zhang H, Zhu M, Qiu Q, Wang Q, Yan X, Kong C, Hao J, Wei C, Tang Y, Qin W, Li Y, Wang F, Guo D, Zhou A, Zuo X, Yu Y, Li D, Zhao L, Jin H, Jia J. PSEN1, PSEN2, and APP mutations in 404 Chinese pedigrees with familial Alzheimer's disease. Alzheimers Dement. 2020 Jan;16(1):178-191. doi: 10.1002/alz.12005. PMID 31914229
- [Result] Qiu Q, Shen L, Jia L, Wang Q, Li F, Li Y, Jia J. A Novel PSEN1 M139L Mutation Found in a Chinese Pedigree with Early-Onset Alzheimer's Disease Increases Abeta42/Abeta40 ratio. J Alzheimers Dis. 2019;69(1):199-212. doi: 10.3233/JAD-181291. PMID 30958370
- [Result] Shen L, Qin W, Wu L, Zhou A, Tang Y, Wang Q, Jia L, Jia J. Two novel presenilin-1 mutations (I249L and P433S) in early onset Chinese Alzheimer's pedigrees and their functional characterization. Biochem Biophys Res Commun. 2019 Aug 13;516(1):264-269. doi: 10.1016/j.bbrc.2019.05.185. Epub 2019 Jun 21. PMID 31235249
- [Result] Qiu Q, Jia L, Wang Q, Zhao L, Jin H, Li T, Quan M, Xu L, Li B, Li Y, Jia J. Identification of a novel PSEN1 Gly111Val missense mutation in a Chinese pedigree with early-onset Alzheimer's disease. Neurobiol Aging. 2020 Jan;85:155.e1-155.e4. doi: 10.1016/j.neurobiolaging.2019.05.018. Epub 2019 May 31. PMID 31235344
- [Result] Li W, Pang Y, Wang Y, Mei F, Guo M, Wei Y, Li X, Qin W, Wang W, Jia L, Jia J. Aberrant palmitoylation caused by a ZDHHC21 mutation contributes to pathophysiology of Alzheimer's disease. BMC Med. 2023 Jun 26;21(1):223. doi: 10.1186/s12916-023-02930-7. PMID 37365538
- [Result] Quan M, Wang Q, Qin W, Wang W, Li F, Zhao T, Li T, Qiu Q, Cao S, Wang S, Wang Y, Jin H, Zhou A, Fang J, Jia L, Jia J. Shared and unique effects of ApoEepsilon4 and pathogenic gene mutation on cognition and imaging in preclinical familial Alzheimer's disease. Alzheimers Res Ther. 2023 Feb 28;15(1):40. doi: 10.1186/s13195-023-01192-y. PMID 36850008
- See also: CFAN Website — http://www.chinacfan.org

DOCUMENTS (1):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT03657732/Prot_000.pdf